CLINICAL TRIAL: NCT03224533
Title: Association Between Walnut Consumption and Diabetes Risk in NHANES May be Gender Sex Specific
Brief Title: Walnut Consumption and Diabetes Risk
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: California Walnut Commission (Other)
Responsible Party: Principal Investigator, Lenore Arab, PhD, Principal Investigator, University of California, Los Angeles
Other Study IDs: WALNUT6DIABETES
Record Dates: First submitted 2017-07-15; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Diabetes Mellitus
Keywords: nut consumption; NHANES; epidemiology; plasma glucose; hemoglobin A1c
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- No Nuts: All other foods that did not include walnuts or other nuts were classified as "no nuts" (NN).
  Interventions: Diagnostic Test: Diabetes Outcome
- Other Nuts: Foods codes describing nuts that are not walnuts (i.e. cashew nuts, pistachios, etc.) or nut-containing foods that do not commonly contain walnuts (e.g. granola) were classified as "other nuts" (ON).
  Interventions: Diagnostic Test: Diabetes Outcome
- Walnuts with other nuts: food codes describing nut mixes and foods that commonly include walnuts were classified as "walnuts with other nuts" (WwON)
  Interventions: Diagnostic Test: Diabetes Outcome
- Walnuts with high certainty: Foods consisting entirely or mostly of walnuts were classified as "walnuts with high certainty" (WwHC)
  Interventions: Diagnostic Test: Diabetes Outcome

INTERVENTIONS:
Diagnostic Test: Diabetes Outcome — based on self report definition, fasting plasma glucose, and hemoglobin A1c

SUMMARY:
Multiple NHANES surveys were combined and weighted to evaluate relationships between walnut consumption and type 2 diabetes mellitus using various independent measures of diabetes status and risk. After risks were ascertained, interactions with gender were analyzed.

DETAILED DESCRIPTION:
Background. Dietary interventions and cohort studies of tree nuts lowering glucose levels for diabetes suggest a possible effect with walnuts. Objective. To examine the associations between walnut consumption and diabetes risk through data from the National Health and Nutrition Examination Survey (NHANES). Methods. NHANES survey data for 1999 through 2014 was pooled for adults with 24 hour recall dietary data. Risk of diabetes was based on self-report, medication use, fasting plasma glucose levels, and hemoglobin A1c (HbA1c) levels. Individuals were characterized as reporting consumption of walnuts, mixed 'nuts', or no nuts.

ELIGIBILITY:
Inclusion Criteria:

* NHANES data from 1999-2014 with food recalls and dietary food intake

Exclusion Criteria:

* not having data on either day of the 24-hour food intake
* individuals who consumed peanuts, but not other nuts on the day of recall, were excluded from the analysis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The National Health and Nutrition Examination Survey (NHANES) is a cross-sectional, probability survey administered to the US civilian population aged from 0 to 85 years. This study used continuous NHANES data collected from 1999 to 2014, covering eight cycles of data collection (N=82,091). Participants were excluded from analysis for being under 18 (N=34,735) and not having data on either day of the 24-hour food intake (N=6,533). In an attempt to have a control group free of nut consumers, individuals who consumed peanuts, but not other nuts on the day of recall, were excluded from the analysis (N=6,702). After exclusions, our analytic sample N was 34,121, representing a population size of approximately 176 million individuals.
Sampling Method: Probability Sample
Enrollment: 34121 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Diabetes Outcome- self report | 1999-2014
  Based on self-report as told by a doctor
Diabetes Outcome- Fasting Plasma Glucose | 1999-2014
  Based on FPG levels
Diabetes Outcome- Hemoglobin A1c | 1999-2014
  Based on HbA1c levels
Diabetes Outcome- Combined Definition | 1999-2014
  Based on both FPG and HbA1c levels

SECONDARY OUTCOMES:
Sex Interaction | 1999-2014
  based on the previously stated definition outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Lenore Arab, MSc, PhD, Principal Investigator — David Geffen School of Medicine
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brennan AM, Sweeney LL, Liu X, Mantzoros CS. Walnut consumption increases satiation but has no effect on insulin resistance or the metabolic profile over a 4-day period. Obesity (Silver Spring). 2010 Jun;18(6):1176-82. doi: 10.1038/oby.2009.409. Epub 2009 Nov 12. PMID 19910942
- [Background] Kalgaonkar S, Almario RU, Gurusinghe D, Garamendi EM, Buchan W, Kim K, Karakas SE. Differential effects of walnuts vs almonds on improving metabolic and endocrine parameters in PCOS. Eur J Clin Nutr. 2011 Mar;65(3):386-93. doi: 10.1038/ejcn.2010.266. Epub 2010 Dec 15. PMID 21157477
- [Background] Katz DL, Davidhi A, Ma Y, Kavak Y, Bifulco L, Njike VY. Effects of walnuts on endothelial function in overweight adults with visceral obesity: a randomized, controlled, crossover trial. J Am Coll Nutr. 2012 Dec;31(6):415-23. doi: 10.1080/07315724.2012.10720468. PMID 23756586
- [Background] Ma Y, Njike VY, Millet J, Dutta S, Doughty K, Treu JA, Katz DL. Effects of walnut consumption on endothelial function in type 2 diabetic subjects: a randomized controlled crossover trial. Diabetes Care. 2010 Feb;33(2):227-32. doi: 10.2337/dc09-1156. Epub 2009 Oct 30. PMID 19880586
- [Background] Mukuddem-Petersen J, Stonehouse Oosthuizen W, Jerling JC, Hanekom SM, White Z. Effects of a high walnut and high cashew nut diet on selected markers of the metabolic syndrome: a controlled feeding trial. Br J Nutr. 2007 Jun;97(6):1144-53. doi: 10.1017/S0007114507682944. Epub 2007 Mar 7. PMID 17381974
- [Background] Tapsell LC, Batterham MJ, Teuss G, Tan SY, Dalton S, Quick CJ, Gillen LJ, Charlton KE. Long-term effects of increased dietary polyunsaturated fat from walnuts on metabolic parameters in type II diabetes. Eur J Clin Nutr. 2009 Aug;63(8):1008-15. doi: 10.1038/ejcn.2009.19. Epub 2009 Apr 8. PMID 19352378
- [Background] Tapsell LC, Gillen LJ, Patch CS, Batterham M, Owen A, Bare M, Kennedy M. Including walnuts in a low-fat/modified-fat diet improves HDL cholesterol-to-total cholesterol ratios in patients with type 2 diabetes. Diabetes Care. 2004 Dec;27(12):2777-83. doi: 10.2337/diacare.27.12.2777. PMID 15562184
- [Background] Wu L, Piotrowski K, Rau T, Waldmann E, Broedl UC, Demmelmair H, Koletzko B, Stark RG, Nagel JM, Mantzoros CS, Parhofer KG. Walnut-enriched diet reduces fasting non-HDL-cholesterol and apolipoprotein B in healthy Caucasian subjects: a randomized controlled cross-over clinical trial. Metabolism. 2014 Mar;63(3):382-91. doi: 10.1016/j.metabol.2013.11.005. Epub 2013 Nov 12. PMID 24360749
- [Background] Moravej H, Salehi A, Razavi Z, Moein MR, Etemadfard H, Karami F, Ghahremani F. Chemical Composition and the Effect of Walnut Hydrosol on Glycemic Control of Patients With Type 1 Diabetes. Int J Endocrinol Metab. 2016 Jan 30;14(1):e34726. doi: 10.5812/ijem.34726. eCollection 2016 Jan. PMID 27335580
- [Background] Bullard KM, Ali MK, Imperatore G, Geiss LS, Saydah SH, Albu JB, Cowie CC, Sohler N, Albright A, Gregg EW. Receipt of Glucose Testing and Performance of Two US Diabetes Screening Guidelines, 2007-2012. PLoS One. 2015 Apr 30;10(4):e0125249. doi: 10.1371/journal.pone.0125249. eCollection 2015. PMID 25928306
- [Background] Guo K, Zhou Z, Jiang Y, Li W, Li Y. Meta-analysis of prospective studies on the effects of nut consumption on hypertension and type 2 diabetes mellitus. J Diabetes. 2015 Mar;7(2):202-12. doi: 10.1111/1753-0407.12173. Epub 2014 Jul 29. PMID 24893671
- [Background] Luo C, Zhang Y, Ding Y, Shan Z, Chen S, Yu M, Hu FB, Liu L. Nut consumption and risk of type 2 diabetes, cardiovascular disease, and all-cause mortality: a systematic review and meta-analysis. Am J Clin Nutr. 2014 Jul;100(1):256-69. doi: 10.3945/ajcn.113.076109. Epub 2014 May 21. PMID 24847854
- [Background] Zhou D, Yu H, He F, Reilly KH, Zhang J, Li S, Zhang T, Wang B, Ding Y, Xi B. Nut consumption in relation to cardiovascular disease risk and type 2 diabetes: a systematic review and meta-analysis of prospective studies. Am J Clin Nutr. 2014 Jul;100(1):270-7. doi: 10.3945/ajcn.113.079152. Epub 2014 May 7. PMID 24808491
- [Background] Pan A, Sun Q, Manson JE, Willett WC, Hu FB. Walnut consumption is associated with lower risk of type 2 diabetes in women. J Nutr. 2013 Apr;143(4):512-8. doi: 10.3945/jn.112.172171. Epub 2013 Feb 20. PMID 23427333
- [Background] Guo F, Moellering DR, Garvey WT. Use of HbA1c for diagnoses of diabetes and prediabetes: comparison with diagnoses based on fasting and 2-hr glucose values and effects of gender, race, and age. Metab Syndr Relat Disord. 2014 Jun;12(5):258-68. doi: 10.1089/met.2013.0128. Epub 2014 Feb 10. PMID 24512556